CLINICAL TRIAL: NCT02950194
Title: Navel Sparing Retro-muscular Mesh Augmentation and Panniculectomy for the Treatment of Post-partum Abdominal Wall Insufficiency (PPAWI)
Brief Title: Mesh Augmentation and Panniculectomy for the Treatment of Post-partum Abdominal Wall Insufficiency
Acronym: PPAWI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Filip Muysoms, surgeon, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: PPAWI
Record Dates: First submitted 2016-10-24; First posted 2016-11-01 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Mesh Augmentation
Keywords: mesh; rectus diastasis; panniculectomy; abdominoplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PPAWI: patients with multidisciplinary PPAWI approach
  Interventions: Procedure: PPAWI

INTERVENTIONS:
Procedure: PPAWI — One-step procedure of a panniculectomy performed by a plastic surgeon together with a mesh augmentation of the abdominal wall by a general surgeon.

SUMMARY:
The aim of this study is to evaluate this multidisciplinary surgical approach of PPAWI (one-step procedure a panniculectomy by a plastic surgeon was performed together with a mesh augmentation of the abdominal wall by a general surgeon) at least 1 year post-operatively. Evaluation of the PPAWI approach by clinical examination with Quality of Life questionnaire and by ultrasound examination.

DETAILED DESCRIPTION:
PPAWI (post partum abdominal wall insufficiency) is an acronym first introduced during Congress of the European Hernia Society in 2013. It is a pathological condition induced by abdominal distension during pregnancy. General laxity of the anterior abdominal wall develops because of diastasis of the rectus abdominis muscles and excess of skin and panniculus. This has important repercussion on abdominal wall function and its aesthetics. This diastasis is induced by abdominal distension and hormonal influences.

To evaluate diastasis of the rectus abdominis the inter-recti distance (IRD) is measured by ultrasound. When it is 3cm or more, it is defined as diastasis of recti abdominis.

An operation is indicated when there is an aesthetic problem and/or the abdominal wall function is impaired e.g. by loss of integrity of myofascial system and altered angle of attachment, which results in loss of abdominal muscle strength and endurance and loss of pelvic stabilization.

Since September 2013, 11 patients underwent an one-step procedure in which a panniculectomy/ abdominoplasty performed by a plastic surgeon was combined by a mesh augmentation of the abdominal wall with a Parietex Progrip Self Fixating Mesh performed by a general surgeon in the Maria Middelares hospital, Ghent, Belgium.

The study will be conducted in the department of surgery in the Maria Middelares hospital, Ghent, Belgium. Dr. Filip Muysoms (general surgeon) selected all patient that have previous been operated together with Dr. Rudolf Vertriest (plastic surgeon) with PPAWI technique. Ultrasound will be performed by Dr. Beckers subsequently pre- and postoperative. Pictures to evaluate the esthetic result will be taken by Dr. Vertriest pre- and postoperative.

The aim of this study is to evaluate this multidisciplinary surgical approach of PPAWI at least one year post-operatively by clinical and radiological examination.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients who underwent an abdominal wall repair and an abdominoplasty in one-step technique

Exclusion Criteria:

* Pregnancy
* No Informed Consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 11 patients were already operated by Dr. Filip Muysoms and Dr. Rudolf Vertriest
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the rectus diastasis by ultrasound | more than 12 months post-operatively
  Evaluation of the rectus diastasis after abdominoplasty with mesh augmentation using ultrasound at least 12 months post-operatively

SECONDARY OUTCOMES:
Aesthetic result | more than 12 months post-operatively
  Aesthetic result evaluated by physical examination
Quality of Life score | more than 12 months post-operatively
  Quality of Life score assessment with the EuraHS QoL score

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD, PhD, Principal Investigator — Maria Middelares hospital; Fien Decuypere, MD, Study Chair — Maria Middelares hospital
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No